CLINICAL TRIAL: NCT02831504
Title: Myotonic Dystrophy Type 1 (DM1) Deep Phenotyping to Improve Delivery of Personalized Medicine and Assist in the Planning, Design and Recruitment of Clinical Trials
Brief Title: PhenoDM1 (Myotonic Dystrophy Type 1 Natural History Study)
Acronym: PhenoDM1
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 7491
Record Dates: First submitted 2016-03-22; First posted 2016-07-13 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Myotonic Dystrophy Type 1
Keywords: Myotonic Dystrophy type 1; DM1; Muscular Dystrophy; Neuromuscular Diseases
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophies; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All blood and urine will be processed and stored in Newcastle Biobank for Research of Neuromuscular Disorders (Newcastle and North Tyneside 1 -REF/08/H0906/28).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myotonic Dystrophy type 1 (DM1) patients: Natural History Study

SUMMARY:
PhenoDM1 will use patient reported outcomes to assess levels of pain, fatigue and quality of life in this cohort. Clinical and functional outcomes will look at muscle wasting and levels of myotonia. DNA, RNA, serum and CSF samples will be taken from all patients so that additional genetic and molecular biomarker analysis can be carried out. A subset of patients will undergo detailed sleep studies along with skeletal muscle MRI of the lower limbs. This study will complement the work of other groups currently looking at myotonic dystrophy type 1 using the same outcomes and measures where possible.

DETAILED DESCRIPTION:
Myotonic Dystrophy type I (DM1) is the most common form of adult muscular dystrophy, affecting 1 in 8000 individuals. It is an autosomal dominant disorder with multisystemic involvement of multiple organs and tissues, namely brain, heart, endocrine system, eyes and both smooth and skeletal muscles. It results from the CTG expansion of an untranslated region 3' terminal of the DMPK gene which causes a disturbance of the RNA metabolism, in particular defective splicing of various pre-mRNAs such as the muscular chloride channel (causing myotonia), the insulin receptor (causing diabetes) and others. We will carry out an in-depth characterisation of 400 adult DM1 patients identified from local clinical populations across England and through the national DM Registry. Over a two year period we will take measurements 12 months apart to address specific symptoms that cause major quality of life impairment including muscle weakness, myotonia, excessive daytime sleepiness and cognitive impairment. DNA samples will be collected in order to determine the CTG repeat length and serum samples for biomarker identification. We will carry out muscle MRI and sleep studies in a subset of 50 patients. The implemented measures will capitalise on the efforts of previous cohort studies ensuring that all measures are comparable with existing datasets.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria

1. 18 years of age or over
2. Genetic confirmation of Myotonic Dystrophy Type 1
3. Able to consent and willing to participate throughout the duration of the study.

Additional Inclusion Criteria for MRI study:

1. Aged between 18 and 55 years
2. Ambulant or ambulant-assisted

Additional Inclusion Criteria for sleep study:

1. Aged between 18 and 55 years

Exclusion Criteria:

Main Exclusion Criteria

1. Inability to give informed consent
2. If the clinician presumes that the patient will not be able to perform any of the motor function tests involved (Six Minute Walk Test, 30 Seconds Sit and Stand Test, Timed 10-Meter Walk Test)
3. Inability to perform the cardiac and pulmonary assessments

Additional Exclusion Criteria for MRI study:

1. Pacemaker, ICD or non-MRI-compatible prosthetic material.

Additional Exclusion Criteria for sleep study:

1. ventilated patients
2. patients medicated with stimulants, including Modafinil
3. patients medicated with benzodiazepines or antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria will be limited to those over 18 years of age, with a genetic confirmation of DM1 who are able to provide informed consent. This unrestrictive approach will enable assessment of a true cross-section of the population, including those with congenital, childhood and adult onset. Two substudies will be open to a subset of patients, one assessing muscle through MRI and on focussing on sleep and fatigue. Additional restrictions may be in place to ensure the safety of the participants during these studies.
  Informed consent will be obtained from all patients, including detailed patient information. Sharing and storage of data and samples will be discussed in this information and covered appropriately in the consent.
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Strength and function | 9-12 months
  These assessments include:
  * Manual Muscle Testing
  * Quantitative Muscle Testing (Hand Held Myometry, Hand-Grip Dynamometry)
  * Pulmonary function testing (FVC and MIP)
  * Functional evaluations (Nine Hole Peg Test, Six Minute Walk Test, 30 Seconds Sit and Stand Test, Timed 10-Meter Walk Test, Scale for Assessment and Rating of Ataxia Scale, Accelerometry Assessment)

SECONDARY OUTCOMES:
Cognitive assessment | 9-12 months
  These questionnaires include:
  * Mini-Mental State Examination (MMS)
  * Trail Making Test (TMT)
  * Apathy Evaluation Scale (AES)
Quality of Life using patient-reported outcomes | 9-12 months
  These questionnaires include:
  * Individualised Neuromuscular Quality Of Life (InQoL)
  * Myotonic Dystrophy Health Index (MDHI)
Fatigue and Daytime Sleepiness assessment using patient-reported outcomes | 9-12 months
  These questionnaires include:
  * Checklist Individual Strength
  * Epworth Sleepiness Scale
  * Fatigue and Daytime Sleepiness Scale
Pain assessment using patient-reported outcomes | 9-12 months
  These questionnaires include:
  * McGill questionnaire
  * IVR Scale
Blood and Urine collection for genetic and molecular biomarker analysis | 9-12 months
  Collection of: RNA, DNA, Serum and Urine
Blood collection for Glycated Haemoglobin (HbA1c), Thyroid hormones, Androgens (in males only) analysis | 9-12 months

OTHER OUTCOMES:
Sleep Study | 9-12 months
  Assessment by polysomnography and maintenance of wakefulness test (MWT)
Skeletal Muscle MRI of the lower extremities | 9-12 months
  Three imaging scans will be acquired of the lower extremities: T1-weighted images, TIRM images and Dixon images.

CONTACTS AND LOCATIONS:
Overall Officials: Hanns Lochmuller, MD, FAAN, Principal Investigator — University of Newcastle Upon-Tyne; Chris Turner, FRCP, PhD, Principal Investigator — National Hospital for Neurology and Neurosurgery
Locations (2):
- United Kingdom (2):
  - Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle upon Tyne, Tyne and Wear
  - University College London Hospitals NHS Foundation Trust, National Hospital for Neurology and Neurosurgery, London

IPD SHARING:
Plan to Share IPD: Yes